CLINICAL TRIAL: NCT00882843
Title: Feasibility Study for the Use of Low-magnitude, High Frequency Mechanical Stimulation of Bone in Persons With SCI
Brief Title: Feasibility Study for the Use of Low-magnitude, High Frequency Mechanical Stimulation of Bone in Persons With Spinal Cord Injury (SCI)
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4162C-9
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Spinal Cord Injuries
Keywords: Vibrating plate; Mechanical Stimulation; Osteoporosis
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Healthy Able bodied Control
- Group 2: Spinal Cord Injury

SUMMARY:
In persons with SCI, because of inherent considerations, the use of mechanical stimulation has not been studied to determine improvement in bone mass. To achieve maximum transmission of the vibration from a vibrating plate to the lower body, the legs must be extended and the feet firmly placed against the surface plate of the device. Thus, these logistical considerations must be addressed to perform this mechanical intervention in persons with SCI. In those with complete or almost complete motor injury, there is lack of musculoskeletal function below the level of the lesion, which would prevent rigid straight leg extension and pressing one's feet against a surface, regardless of the angle of tilt that would permit adequate transmission of impulse in an able-bodied individual (preliminary data). However, in one subject with SCI, there was measurable, albeit low level, transmission of vibration with increasing angles of tilt (preliminary data). Because of the ability to transmit some signal in an individual with complete SCI, the possibility exists that with forms or mechanical support/manipulation, greater signal transmission may be possible. The study will be able to determine the best angle to transmit mechanical vibration through the lower body of SCI patients.

DETAILED DESCRIPTION:
Experiments will be performed in 12 persons with SCI and 10 healthy able-bodied to optimize the methodology for transmission of the mechanical impulse to the lower extremities in persons with SCI. This will entail the following combinations:

1. positional modification (sitting, lying or standing if tolerable);
2. bracing the knee to prevent flexion/extension;
3. bracing the legs above and/or below the knee;
4. supporting the ankle;
5. tilting the surface (tilt table) to a maximum angle of 45 degrees;
6. Standing with the assistance of a standing frame if subject can tolerate standing for 5 minute time periods.
7. increasing the magnitude of the plate acceleration (0.2-0.6g); and
8. mechanically pressing the legs (ankle and knee joints relatively fixed in position by an orthotic device) against the plate by a spring-loaded method (it is envisioned that a padded belt-like article will be worn around the waist and would be attached with bungee cords (or springs) to each side of the vibrating plate; the maximum force delivered would be equal to 50 lbs or one-third of total body weight, whichever is less).

An accelerometer for the measurement of impulse generation will be placed on the surface of the vibrating plate between the feet; a second will be placed on the shin about 4 inches below the knee (attached with double sided tape and athletic bandage wrap); a third accelerometer will be placed in the mouth as a bite-bar. Measurements would be acquired with combinations of body position, joint/leg fixation, magnitude of plate acceleration ("g" force), and mechanical force pressing the feet against the plate to determine the optimal transmission of impulse.

This study will determine the optimal of the methodology for using the vibrating plate to transmit an impulse in persons with chronic SCI, with the anticipation of its application to increase bone mass in individuals with acute or chronic SCI. It is anticipated that each session will be between 30 and 120 minutes. An individual may voluntarily participate in as many as 5 sessions. The knowledge gained from the first sets of studies will obviate the need to perform less effective methods of mechanical signal transmission in subsequent studies. It is anticipated that once the most effective, as well as clinically applicable, form of mechanical stimulation is identified, it will be performed in most of the subjects. This preliminary study will also provide the information required to determine practical aspects of the length of each session and number of sessions per week in a future intervention trial.

Since this research may have adverse effects on an unborn child and should not be done during pregnancy, we will administer a pregnancy test when appropriate. Subjects will be asked to avoid becoming pregnant and use contraceptives, take precautions against becoming pregnant.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic spinal cord injury or healthy able-bodied
2. 18+ years of age

Exclusion Criteria:

1. Severe underlying chronic illness (cardiac, pulmonary, gastrointestinal, etc.)
2. Flexion contractures of the lower extremities
3. Femur or tibia fracture or history of extensive bone trauma
4. History of prior bone disease
5. Post-menopausal women
6. Renal disease (creatinine clearance < 40 ml/min)
7. Endocrine disorders known to be associated with osteoporosis (hyperthyroidism, hypercortisolism, hypogonadism)
8. Alcoholism
9. Seizure disorders
10. All pressure ulcers of the sacral/pelvic region, lower extremities, and heels
11. Pacemakers, implanted cardiac defibrillators, or any other electrical cardiac device
12. Implanted rods placed between 2 or more vertebral segments
13. Pregnant women (pregnancy test will be administered when applicable)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ten ambulatory able-bodied and Twelve non-ambulatory subjects with SCI will be enrolled to participate
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Experiments will be to optimize the methodology for transmission of the mechanical impulse to the lower extremities in persons with SCI. | one day

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States